CLINICAL TRIAL: NCT07101614
Title: An Open-label, Randomized, Multi-center, Multi-cohort Clinical Study of JS004 and Toripalimab Combined With Chemotherapy vs Toripalimab Combined With Chemotherapy vs Chemotherapy Alone as Neoadjuvant Therapy for Stage II-III Triple-negative Breast Cancer (TNBC).
Brief Title: A Randomized Study of JS004 and Toripalimab Combined With Chemotherapy vs Toripalimab Combined With Chemotherapy vs Chemotherapy Alone as Neoadjuvant Therapy for Stage II-III Triple-negative Breast Cancer (TNBC).
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Shengjing Hospital, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNBC-IIT-JS004-N01
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: TNBC - Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — toripalimab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- JS004+Toripalimab+chemotherapy (Experimental)
  Interventions: Drug: JS004 in combination with toripalimab and chemotherapy
- Toripalimab+chemotherapy (Experimental)
  Interventions: Drug: Toripalimab and chemotherapy
- chemotherapy (Other)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: JS004 in combination with toripalimab and chemotherapy — BTLA inhibitor (JS004):200mg, IV infusion , d1, Q3W;(1-24 week)
  Toripalimab:240mg, IV infusion , d1, Q3W;(1-24 week)
  Carboplatin: IV infusion,AUC=5, d1,q3w(OR AUC=1.5,d1,qw);(1-12 week)
  Paclitaxel:IV infusion,80 mg/m2,qw;(1-12 week)
  Doxorubicin:IV infusion,60 mg/m2,q3w(OR Epirubicin:IV infusion,90 mg/m2,q3w);(13-24 week)
  Cyclophosphamide:IV infusion,600 mg/m2,q3w(13-24 week)
  Arms: JS004+Toripalimab+chemotherapy
Drug: Toripalimab and chemotherapy — Toripalimab:240mg, IV infusion , d1, Q3W;(1-24 week)
  Carboplatin: IV infusion,AUC=5, d1,q3w(OR AUC=1.5,d1,qw);(1-12 week)
  Paclitaxel:IV infusion,80 mg/m2,qw;(1-12 week)
  Doxorubicin:IV infusion,60 mg/m2,q3w(OR Epirubicin:IV infusion,90 mg/m2,q3w);(13-24 week)
  Cyclophosphamide:IV infusion,600 mg/m2,q3w(13-24 week)
  Arms: Toripalimab+chemotherapy
Drug: Chemotherapy — Carboplatin: IV infusion,AUC=5, d1,q3w(OR AUC=1.5,d1,qw);(1-12 week)
  Paclitaxel:IV infusion,80 mg/m2,qw;(1-12 week)
  Doxorubicin:IV infusion,60 mg/m2,q3w(OR Epirubicin:IV infusion,90 mg/m2,q3w);(13-24 week)
  Cyclophosphamide:IV infusion,600 mg/m2,q3w(13-24 week)
  Arms: chemotherapy

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of chemotherapy plus toripalimab, with or without JS004,as neoadjuvant therapy for patients with triple-negative breast cancer (TNBC). TNBC patients were randomly assigned in a 2:2:1 ratio to receive either JS004 plus toripalimab plus chemotherapy, toripalimab plus chemotherapy, or chemotherapy alone.Surgery will be performed within 5 weeks after the last dose of neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily participate in this study, sign the informed consent form, demonstrate good compliance, and cooperate with follow-up visits.
2. Age ≥ 18 years.
3. ECOG score ≤ 1.
4. Newly diagnosed, non-metastatic breast cancer of stage II-III, confirmed by histopathology or cytopathology (T1c-2 cN1-2 (≥2cm) or T3-4 cN0-2).
5. Pathologically confirmed hormone receptor-negative (ER and PR negative) and HER2-negative advanced breast cancer. In cases of multiple pathological results, the definition of triple-negative breast cancer is based on the final molecular subtype result from the last biopsy pathology. (ER negativity: immunohistochemical staining in <1% of tumor cells; PR negativity: immunohistochemical staining in <1% of tumor cells; HER2 negativity: immunohistochemical score of 0, 1+, or FISH/CISH negative).
6. Have at least one measurable lesion according to the RECIST v1.1 criteria.
7. Functional levels of vital organs must meet the following requirements (without any corrective treatment with blood components or cytokine growth factors within 14 days before the first dose):

   1. Bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, hemoglobin ≥ 90 g/L.
   2. Liver and kidney function: Albumin level ≥ 3.0 g/dL, total bilirubin ≤ 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN, alkaline phosphatase ≤ 2.5 × ULN, urea nitrogen and serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min (calculated according to the Cockcroft-Gault formula).
   3. Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
   4. Echocardiography (ECHO) showing left ventricular ejection fraction (LVEF) ≥ 50%.
   5. QTcF ≤ 470 msec.
8. Within 7 days before the first dose, women of reproductive potential must have a negative serum pregnancy test and agree to use effective contraceptive measures during the study drug administration and for 6 months after the last dose. For this protocol, women of reproductive potential are defined as sexually mature women who: 1) have not undergone hysterectomy or bilateral oophorectomy, and 2) have not experienced spontaneous menstruation cessation for a continuous period of 24 months (amenorrhea following cancer treatment does not exclude fertility) (i.e., menstruation has occurred at any time within the previous 24 consecutive months). For male patients with female partners of reproductive potential, they must agree to use effective contraceptive measures during the study drug administration and for 6 months after the last dose.
9. Voluntarily participate in this study, sign the informed consent form, demonstrate good compliance, and be willing to cooperate with visits and study-related procedures.

Exclusion Criteria:

1. Prior exposure to drugs targeting the same therapeutic target as the study treatment drug planned for administration.
2. Radiotherapy, chemotherapy, surgery, or other targeted immunotherapy for triple-negative breast cancer before enrollment.
3. Uncontrolled central nervous system metastases (symptomatic or requiring glucocorticoids or mannitol for symptom control).
4. Inflammatory breast cancer, bilateral breast cancer, or occult breast cancer.
5. History of clinically significant or uncontrolled cardiac disease within 6 months before the first dose, including congestive heart failure, angina pectoris, myocardial infarction, or ventricular arrhythmias.
6. Presence of severe concomitant diseases that, in the investigator's judgment, pose a significant risk to the patient's safety or ability to complete the study (including but not limited to severe hypertension not controlled by medication, severe diabetes, active infections, etc.).
7. Malignancy within 5 years before the first dose (except for cured basal cell carcinoma of the skin and cervical carcinoma in situ).
8. Active autoimmune diseases requiring systemic treatment within 2 years before the first dose, except for vitiligo, type 1 diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis requiring only hormone replacement therapy.
9. Receipt of live or attenuated vaccines within 4 weeks before the first dose of the study drug.
10. Known or suspected interstitial pneumonia. Presence of other moderate to severe respiratory diseases within 3 months before the first dose that may interfere with the detection or management of drug-related lung toxicity, including but not limited to idiopathic pulmonary fibrosis, organizing pneumonia/bronchiolitis obliterans, pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease (COPD), obstructive/restrictive lung diseases, etc.; as well as any autoimmune, connective tissue, or inflammatory diseases affecting the lungs, such as rheumatoid arthritis, Sjögren's syndrome, sarcoidosis, etc., or prior total lung resection surgery.
11. Known history of human immunodeficiency virus (HIV) infection.
12. Known history of hepatitis B or active hepatitis C virus infection.
13. Prior allergy to any component or excipient of the study drug planned for administration.
14. Other conditions deemed unsuitable for participation in the study by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate | Up to 30 months
  PCR rate is defined as the proportion of participants who have achieved pathologic complete response (on routine hematoxylin and eosin staining, no tumor cell can be found in tumor bed or lymph node) in all participants.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 30 months
  ORR is defined according to the RECIST v1.1 criteria.
Breast pathologic complete response (bpCR) | Up to 30 months
  The bpCR is defined as the histological evidence of no malignancy in the primary lesion of breast cancer, or only carcinoma in situ (i.e., ypT0/Tis, in accordance with current AJCC staging system).
Residual Cancer Burden (RCB) 0-1 | Up to 30 months
  Rate of RCB 0-1 at time of surgery
Event-free Survival (EFS) | Up to 30 months
  Event free survival (EFS) is defined as the time from randomization to first EFS event. For subjects who had breast cancer surgery, EFS events were post-surgery breast cancer relapse, second primary malignancy or death without recurrence. For subjects who did not have breast cancer surgery, EFS events were death during clinical follow-up or non-completion of any neoadjuvant investigational product due to disease progression
Incidence of adverse event | Up to 30 months
  Including type, incidence, severity, time and so on of adverse events

IPD SHARING:
Plan to Share IPD: No